CLINICAL TRIAL: NCT03510273
Title: Evaluation of the Liger Medical Thermocoagulator for Treatment of Cervical Intraepithelial Lesions in Honduras
Brief Title: Honduras Liger Thermocoagulator Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PATH (Other)
Collaborators: Ashonplafa (Other); Ministry of Health, Honduras (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1018287
Record Dates: First submitted 2018-04-17; First posted 2018-04-27 (Actual); Results first posted 2020-03-06 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2019-10

CONDITIONS: Cervix Cancer; Cervix Lesion
Keywords: Thermocoagulation; Treatment; Cervical precancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia

STUDY DESIGN:
Intervention Model Description: Thermal coagulator ablation treatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Thermocoagulation treatment (Other): Acceptability of Liger Medical Thermocoagulator treatment
  Interventions: Device: Liger Medical Thermocoagulator

INTERVENTIONS:
Device: Liger Medical Thermocoagulator — Thermocoagulation treatment by Liger Medical device (US FDA "510K" clearance received)

SUMMARY:
This was a prospective study to evaluate the short-term safety and acceptability of the Liger Medical thermal coagulation device for treatment of cervical precancerous lesions. Study results will inform the Honduras Ministry of Health regarding potential use of the Liger device for precancer treatment in Honduras and results may be of interest to other Latin American settings as well.

The research was conducted in the Tegucigalpa Region in Honduras in 4 health facilities in urban and peri-urban settings. Participants were women ages 30-49 who met the study eligibility criteria. Human papilloma virus (HPV) and visual inspection with acetic acid (VIA)-positive women who were eligible for ablative treatment were offered thermal coagulation with the Liger instrument to treat their lesions and asked about acceptability of the treatment. At this visit, biopsies were also be taken. Women were followed-up at 1 month to evaluate short-term safety outcomes with a physical exam and receive their biopsy results. Depending on their biopsy results, they will be asked to return for repeat screening, referred for further treatment or asked to come back for a 12-month study visit. At the 12-month visit after treatment, women were followed up to evaluate cure rates.

A second investigational device, Pocket Colposcope, was used to take cervix photos at the enrollment and 12-month study visit with participant consent. The photos were used to explore factors influencing treatment failure. De-identified photos and women's diagnosis information were also shared with the device developers, Duke University, for the purposes of improving their device. Women had the option to opt out of having cervix photos taken and still participate in the treatment portion of the study.

ELIGIBILITY:
Inclusion Criteria:

Women

* Aged 30 to 49 years.
* HPV and VIA positive.
* Eligible for ablative treatment using World Health Organization Guidelines [29].

  * The lesion covers <75% of the cervix, the lesion does not enter the endocervical canal, the entire lesion can be visualized and covered by the Liger Medical Thermocoagulator probe, and there is no suspicion for invasive cancer.

Exclusion Criteria:

* Are pregnant or less than 3 months post-partum
* Are not HPV and VIA positive
* Do not have a cervical lesion that qualifies for ablative treatment
* Have a bleeding disorder or taking anti-coagulant medication.
* Do not give informed consent; or unable to provide the consent.

Ages: 30 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 320 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia de Sanjose, MD, PhD, Principal Investigator — PATH
Locations (1):
- PATH, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One woman was positive for visual inspection with acetic acid, but after enrollment was found to not have documentation of her human papillomavirus test or test result. Therefore, 320 were enrolled but only 319 participated in the study.
Groups:
- Thermocoagulation Treatment: Received thermal coagulation treatment for cervical precancer.
Period: Overall Study
Arm/Group | Thermocoagulation Treatment
Started | 319
Treated With Thermal Coagulation | 319
Completed 1-mth Follow-up Visit & Exited (Completed one-month follow-up visit and exited study per protocol) | 192
Completed 1-mth Follow-up Visit & Cont'd (Completed one-month follow-up visit and continued in study for secondary outcomes) | 126
Completed All One-year Follow up Visits | 118
Completed | 310
Not Completed | 9
Not completed — Withdrawal by Subject | 2
Not completed — Care outside study, ineligible to cont. | 3
Not completed — Moved away from study area | 4

BASELINE CHARACTERISTICS:
Population: No differences from the assignment in the Participant Flow section.
Arm/Group | Thermocoagulation Treatment
Number analyzed (Participants) | 319
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 319
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 319
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Honduras | 319

OUTCOME MEASURES:

1. Primary Outcome: Short-term Safety Concerns for Ablative Treatment
Description: Reported a short-term adverse event. Note: Participants could report more than one discomfort or problem experienced.
Time Frame: 1 month after treatment
Population: All participants were included. Note: Participants could report more than one discomfort or problem experienced.
Measure: Number; unit: participants
Arm/Group | Thermocoagulation Treatment
Number analyzed (Participants) | 319
participants
  Colorless watery discharge | 288
  Brown/black discharge | 106
  Foul-smelling, pus-colored discharge | 100
  Bleeding | 31
  Pain while urinating | 2
  Severe lower abdominal pain | 11
  Fever | 0

2. Primary Outcome: Acceptability of Treatment by Women
Description: Level of pain women experienced during the thermal coagulation procedure will be calculated by the number and percent of women indicating minimal to worst possible levels of pain using the Wong-Baker FACES® pain rating scale. Women's acceptability will also be assessed by asking if they would recommend the Liger Thermocoagulator treatment to a friend or relative who needed similar treatment as well as reasons for her response.
  Wong-Baker FACES® pain rating scale:
  MINIMUM value: 0 (no hurt = best outcome) Value: 2 (hurts little bit) Value: 4 (hurts little more) Value: 6 (hurts even more) Value: 8 (hurts lot more) MAXIMUM value: 10 (hurts whole lot = worst outcome)
Time Frame: Immediately after treatment
Population: Not applicable; all participants were included.
Measure: Count of Participants; unit: Participants
Arm/Group | Thermocoagulation Treatment
Number analyzed (Participants) | 319
Participants
  FACES® level of pain: 0 - no hurt | 62
  FACES® level of pain: 2 - hurts little bit | 168
  FACES® level of pain: 4 - hurts little more | 43
  FACES® level of pain: 6 - hurts even more | 30
  FACES® level of pain: 8 - hurts whole lot | 15
  FACES® level of pain: 10 - hurts worst | 1
  Would recommend treatment to friend/relative | 319
  Would not recommend treatment to friend/relative | 0

3. Secondary Outcome: Percentage of Participants With no Evidence of CIN2-3 Lesions 12 Months After Thermal Coagulation
Description: Percentage of participants with no evidence of cervical intraepithelial neoplasia grade 2 or grade 3 (CIN2-3) at 12 months, based on histological evaluation following the standard criteria from WHO Classification of Tumours, 5th Edition, Volume 4: Female Genital Tumours.
Time Frame: One time, 12 months after treatment
Measure: Number (95% Confidence Interval); unit: % participants
Groups:
- CIN2-3 at Baseline: Biopsy positive at baseline
- < CIN2 at Baseline: Biopsy negative at baseline
Arm/Group | CIN2-3 at Baseline | < CIN2 at Baseline
Number analyzed (Participants) | 69 | 49
% participants | 91.30 [81.7 to 96.1] | 97.96 [86.4 to 99.7]

4. Secondary Outcome: Treatment Failure
Description: Qualitative analysis of cervical photos by an expert colposcopist to explore factors associated with treatment failure, compared characteristics of the cervix and precancerous lesions among women with CIN2-3 at Visit 1 (enrollment) in women whose treatment resulted in lesion disappearance (<CIN2), and women with persistent lesions (CIN2-3) at 12 months. Adequacy of the image included focus, blur, and capture; a well focused image without obstructions (blood, cysts) that captured the whole ectocervix and cervical os was considered adequate. For squamous columnar junction and transformation zone (TZ) visibility, TZ1 signifies a fully visible TZ, TZ2 signifies the TZ or visible lesions extend into the cervical canal and the TZ covers more than 75% of the ectocervix, and TZ3 signifies that the TZ is not at all visible, in accordance with WHO recommendations. Baseline histology reports histological evaluation of lesions as cervical intraepithelial neoplasia grade 2 (CIN2) or 3 (CIN3).
Time Frame: Once, 12 months after treatment
Measure: Count of Participants; unit: Participants
Groups:
- Evidence of Treatment Failure: Women with CIN2-3 at baseline and CIN2-3 at 12 months
- No Evidence of Treatment Failure: Women with CIN2-3 at baseline and <CIN2 at 12 months
Arm/Group | Evidence of Treatment Failure | No Evidence of Treatment Failure
Number analyzed (Participants) | 5 | 63
Participants
  Baseline photo: Adequate | 2 | 38
  Baseline photo: Inadequate | 3 | 25
  Squamous columnar junction visibility: TZ1 | 1 | 20
  Squamous columnar junction visibility: TZ2 | 1 | 4
  Squamous columnar junction visibility: TZ3 | 2 | 39
  Squamous columnar junction visibility: Missing | 1 | 0
  Visible abnormal areas: 0 | 1 | 8
  Visible abnormal areas: 1 | 1 | 23
  Visible abnormal areas: 2+ | 1 | 29
  Visible abnormal areas: Not evaluable | 0 | 2
  Visible abnormal areas: Missing | 2 | 1
  Location of the lesion: Inside the TZ | 4 | 43
  Location of the lesion: Outside the TZ | 0 | 10
  Location of the lesion: Not evaluable | 1 | 10
  Mosaic of the worst lesion: Fine | 0 | 2
  Mosaic of the worst lesion: Coarse | 2 | 7
  Mosaic of the worst lesion: No mosaic | 3 | 50
  Mosaic of the worst lesion: Not evaluable | 0 | 4
  Border of the worst lesion: Irregular | 0 | 10
  Border of the worst lesion: Sharp | 4 | 36
  Border of the worst lesion: Not evaluable | 1 | 17
  Possible diagnosis: No lesion | 1 | 12
  Possible diagnosis: LSIL | 0 | 8
  Possible diagnosis: HSIL | 3 | 25
  Possible diagnosis: Invasion | 1 | 15
  Possible diagnosis: Not evaluable | 0 | 3
  Baseline histology: CIN2 | 3 | 32
  Baseline histology: CIN3 | 2 | 31
  Size of worst lesion (% coverage): 0-4 | 1 | 7
  Size of worst lesion (% coverage): 5-50 | 2 | 38
  Size of worst lesion (% coverage): >50 | 2 | 18
Statistical Analysis 1: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of statistical test: Independence Description: Adequacy of baseline image; p = 0.396, Fisher Exact
Statistical Analysis 2: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of statistical test: Independence Description: Squamous columnar junction visibility; p = 0.351, Fisher Exact
Statistical Analysis 3: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of statistical test: Independence Description: Visible abnormal areas; p = 0.774, Fisher Exact
Statistical Analysis 4: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of statistical test: Independence Description: Location of the lesion; p = 1, Fisher Exact
Statistical Analysis 5: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of statistical test: Independence Description: Mosaic of the worst lesion; p = 0.36, Fisher Exact
Statistical Analysis 6: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of Statistical Test: Independence Description: Acetowhite changes; p = 0.881, Fisher Exact
Statistical Analysis 7: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of Statistical Test: Independence Description: Border of the worst lesion; p = 0.829, Fisher Exact
Statistical Analysis 8: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of Statistical Test: Independence Description: Possible diagnosis; p = 1, Fisher Exact
Statistical Analysis 9: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of Statistical Test: Independence Description: Baseline histology; p = 1, Fisher Exact
Statistical Analysis 10: Comparison: Evidence of Treatment Failure vs No Evidence of Treatment Failure; Test type: Other — Type of Statistical Test: Independence Description: Size of the worst lesion (% coverage); p = 0.493, Fisher Exact

ADVERSE EVENTS:
Time Frame: Between 1 day and 12 months+1 day, depending on when the patient exited the study for any reason.
Description: Self-reported patient data
Arm/Group | Thermocoagulation Treatment
All-Cause Mortality (participants affected / at risk) | 0/319
Serious Adverse Events (participants affected / at risk) | 0/319
Other Adverse Events (participants affected / at risk) | 308/319
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thermocoagulation Treatment (N=319)
High pain during procedure (Reproductive system and breast disorders) | 16 (16)
Mild bleeding/spotting during procedure (not requiring medical attention) (Reproductive system and breast disorders) | 32 (32)
Mild cramping during procedure (not requiring medical attention) (Reproductive system and breast disorders) | 24 (24)
Dizziness during procedure (not requiring medical attention) (General disorders) | 16 (16)
Colorless water discharge within 30 days of procedure (not requiring medical attention) (Reproductive system and breast disorders) | 288 (288)
Brown/black discharge within 30 days of procedure (not requiring medical attention) (Reproductive system and breast disorders) | 106 (106)
Foul smelling, pus colored discharge within 30 days of procedure (not requiring medical attention) (Reproductive system and breast disorders) | 100 (100)
Bleeding within 30 days of procedure (not requiring medical attention) (Reproductive system and breast disorders) | 31 (31)
Attended health facility or saw health provider because of problems. (Reproductive system and breast disorders) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT03510273/Prot_SAP_000.pdf